CLINICAL TRIAL: NCT05414396
Title: Reducing Cancer and Chronic Disease Risk in Underserved Communities: Eat, Move, Live Program
Brief Title: Eat, Move, Live Program for the Reduction of Cancer and Chronic Disease Risk in Underserved Communities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17410; NCI-2022-00180 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17410 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-06-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus; Obesity-Related Malignant Neoplasm
MeSH Terms: conditions — Diabetes Mellitus | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (EML program) (Experimental): Participants attend EML program sessions weekly for 12 weeks including an educational session chronic disease risk reduction via nutrition and physical activity, a physical activity session, and a cooking/taste test demonstration.
  Interventions: Behavioral: Behavioral Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Attend EML program sessions
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests the Eat, Move, Live (EML) Program in reducing the risk of chronic diseases among underserved communities by improving healthy lifestyle practices, increasing physical activity and encouraging healthy eating behaviors. EML is a series of free culturally and linguistically appropriate nutrition and physical activity sessions. The interactive education segment of the EML Program is culturally responsive, and based on the community EML program, and topics will include: nutrition guidelines, reading food labels, recipe modification and healthy food preparation, eating healthy on a budget, chronic diseases information and prevention strategies. The EML program may help reduce the risk of cancer and chronic diseases by encouraging more physical activity and healthy eating behaviors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate program by assessing in combination with standard of care metformin: Changes in participants' knowledge, attitudes, and behavior.

II. To evaluate program by assessing in combination with standard of care metformin: Changes in body measurements.

III. To evaluate program by assessing in combination with standard of care metformin: Changes in biomarkers.

OUTLINE:

Participants attend EML program sessions weekly for 12 weeks including an educational session chronic disease risk reduction via nutrition and physical activity, a physical activity session, and a cooking/taste test demonstration.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to group consent at week 1
* Age over 18
* Able to speak and understand English and/or Spanish

Exclusion Criteria:

* Don't agree to group consent at week 1
* Age younger than 18
* Not able to speak and understand English and/or Spanish
* Can't participate in physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Changes in attitudes and beliefs as measured by questionnaires from baseline to week 12 | Baseline and week 12
  Attitudes and beliefs regarding causes of diabetes asked in questionnaire, measured by endorsing one of the Likert-type scale values ranging from 1 (Agree) to 7 (Disagree).
Changes in behavior as measured by questionnaires from baseline to week 12 | Baseline and week 12
  Behaviors related to food consumption asked in questionnaires, measured by endorsing one of "None", "1", "2-3", "4-6", "7 or more".
Changes in height from baseline to week 12 | Baseline to 12 weeks
  Height measured in meters
Changes in weight from baseline to week 12 | Baseline to 12 weeks
  Weight measured in Kilograms
Changes in waist circumference from baseline to week 12 | Baseline to 12 weeks
  Hip circumference measured in centimeters
Changes in chest circumference from baseline to week 12 | Baseline to 12 weeks
  Chest circumference measured in centimeters
Changes in right upper arm circumference from baseline to week 12 | Baseline to 12 weeks
  Right upper arm circumference measured in centimeters
Changes in left upper arm circumference from baseline to week 12 | Baseline to 12 weeks
  Left upper arm circumference measured in centimeters
Changes in right upper thigh circumference from baseline to week 12 | Baseline to 12 weeks
  Right upper thigh circumference measured in centimeters
Changes in left upper thigh circumference from baseline to week 12 | Baseline to 12 weeks
  Left upper thigh circumference measured in centimeters
Changes in body fat percentage from baseline to week 12 | Baseline to 12 weeks
  Body fat percentage measured in percent using a handheld BMI machine that calculates body fat percentage.
Changes in systolic blood pressure from baseline to week 12 | Baseline to 12 weeks
  Systolic blood pressure measured in mmHG
Changes in diastolic blood pressure from baseline to week 12 | Baseline to 12 weeks
  Diastolic blood pressure measured in mmHG
Changes in hip circumference from baseline to week 12 | Baseline to 12 weeks
  Hip circumference measured in centimeters
Changes in biomarkers | Baseline to 12 weeks
  Will be collected at baseline and follow up based on glycosylated hemoglobin (A1C) measuring guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria L Seewaldt, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States